CLINICAL TRIAL: NCT03417466
Title: A Pivotal Study to Evaluate Enlite™ Sensor Performance With iPro™2 in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP313
Record Dates: First submitted 2018-01-25; First posted 2018-01-31 (Actual); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Type I Type II
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Study arm (Experimental): Use Enlite Sensor over 144 hours (6 days) when inserted in the abdomen and used with the iPro2 and undergo one Yellow Springs Instrument (YSI™) frequent sample testing (FST) (Day 1, 3-4, or 6).
  Interventions: Device: Enlite 1 connected to iPro2 recorder

INTERVENTIONS:
Device: Enlite 1 connected to iPro2 recorder — Use Enlite Sensor over 144 hours (6 days) when inserted in the abdomen and used with the iPro2 in subjects age 14 - 75 years.

SUMMARY:
The purpose of this study is to demonstrate the performance and safety of the Enlite Sensor over 144 hours (6 days) when inserted in the abdomen and used with the iPro2 in subjects age 14 - 75 years.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, prospective single-sample correlational design without controls. Up to 72 subjects will be enrolled in order to have approximately 60 subjects complete the study. Three investigational centers in China will be used during this study.

Each subject will wear the following devices:

• Two Enlite Sensors each connected to an iPro2 for approximately 6 days

Sensor Location:

• The 2 Enlite Sensors will be worn in the abdomen area. Investigational center staff will insert sensors and connect to the iPro2s.

During the study, each subject will be randomized and undergo one Yellow Springs Instrument (YSI™) frequent sample testing (FST) (Day 1, 3-4, or 6).

During the study, subjects will continue with their current diabetes regimen independent of the study devices. Subjects will be instructed by the investigational center that they are not to use the study devices (except for the study meter) for the management of their diabetes. The Study Meter may be used for treatment decisions and calibration of Enlite Sensor.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 14 - 75 years of age at time of screening
2. Subject has a clinical diagnosis of type 1 or 2 diabetes as determined via medical record or source documentation by an individual qualified to make a medical diagnosis
3. Subject has adequate venous access as assessed by investigator or appropriate staff
4. Subject is willing to follow the study procedures and willing to come to study visits.
5. Subject is willing to perform at least 4 self-monitoring of blood glucose (SMBG) per day for 6 days

Exclusion Criteria:

1. Subject will not tolerate tape adhesive in the area of Enlite Sensor placement as assessed by qualified individual.
2. Subject has any unresolved adverse skin condition in the area of study device or device placement (e.g., psoriasis, rash, Staphylococcus infection)
3. Subject is actively participating in an investigational study (drug or device) wherein they have received treatment from an investigational study (drug or device) in the last 2 weeks
4. Subject is female and has a positive pregnancy screening test
5. Females of child bearing age and who are sexually active should be excluded if they are not using a form of contraception deemed reliable by investigator
6. Subject is female and plans to become pregnant during the course of the study
7. Subject has a hematocrit (Hct) lower than the normal reference range
8. Subject may not be on the research staff of those performing this study

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, MD, Principal Investigator — Shanghai 6th People's Hospital; Xiaofeng Lv, MD, Principal Investigator — PLA Army General Hospital; Hong Li, MD, Principal Investigator — Sir Run Run Shaw Hospital
Locations (3):
- China (3):
  - PLA Army General Hospital, Beijing
  - Sir Run Run Shaw Hospital School of Medicine Zhejiang University, Hangzhou
  - Shanghai Sixth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 72 subjects signed the informed consent form and completed the screening. Five subjects failed the screening. One subject withdrew before wearing the sensor.
Period: Overall Study
Arm/Group | Study Arm
Started | 66
Completed | 66
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Arm
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.82 (12.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 66
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 66

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage of Enlite Sensor Values That Are Within 20% Agreement of Gold Standard (Yellow Springs Instrument (YSI) YSI Plasma Glucose Values)
Description: Primary endpoint is the mean percentage of Enlite Sensor Values from primary sensor that are within 20% agreement of YSI plasma glucose values (within 20 mg/dL if YSI <= 80 mg/dL) during YSI frequent sampling testing (FST) days.
Time Frame: YSI FST days (Day 1, 3-4, or 6 of sensor wear)
Population: Subjects who have Enlite sensor inserted and have at least one paired Enlite sensor and YSI measurement. 66 subjects have Enlite sensor inserted, of which one subject has no paired Enlite sensor and YSI measurement.
Measure: Mean (Standard Deviation); unit: percentage of paired readings
Arm/Group | Study Arm
Number analyzed (Participants) | 65
percentage of paired readings | 85.74 (22.26)

2. Secondary Outcome: Enlite Sensor Accuracy Mean Absolute Relative Difference (MARD)
Description: Enlite sensor values from primary sensor were compared to YSI plasma glucose values during YSI FST days (Day 1, 3-4, or 6). MARD = Mean of ((Absolute difference of YSI reference and Sensor glucose values / YSI reference glucose values) * 100). Therefore, the unit of MARD is percentage (%).
Time Frame: YSI FST days (Day 1, 3-4, or 6 of sensor wear)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of difference
Arm/Group | Study Arm
Number analyzed (Participants) | 65
percentage of difference | 10.11 (8.16)

3. Secondary Outcome: Clarke Error Grid Analysis of Paired Sensor and YSI Plasma Glucose Values
Description: Clarke Error Grid compared the paired primary sensor and YSI reference glucose values. Zone A represents a region where sensor values that are within 20% of YSI reference values, or both sensor and YSI reference values are less than 70 mg/dL. Values in Zone A are "clinically accurate in that they would lead to clinically correct treatment decisions". Zone B represents sensor values that deviate YSI reference values by more than 20%, but "would lead to benign or no treatment". Ideal situation is 100% in Zone A + B.
Time Frame: YSI FST days (Day 1, 3-4, or 6 of sensor wear)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of paired readings
Arm/Group | Study Arm
Number analyzed (Participants) | 65
percentage of paired readings | 98.4 [97.8 to 99.0]

4. Secondary Outcome: Consensus Error Grid Analysis of Paired Sensor and YSI Plasma Glucose Values
Description: Consensus Error Grid (or Parkes error grid) compared the paired primary sensor and YSI reference glucose values. Zone A is defined in the Parkes error grid as the zone of "clinical accurate measurements with no effect on clinical action", Zone B as "altered clinical action with little or no effect on clinical outcome". Ideal situation is 100% in Zone A + B.
Time Frame: YSI FST days (Day 1, 3-4, or 6 of sensor wear)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of paired readings
Arm/Group | Study Arm
Number analyzed (Participants) | 65
percentage of paired readings | 99.4 [99.0 to 99.8]

ADVERSE EVENTS:
Time Frame: 6 days
Arm/Group | Study Arm
All-Cause Mortality (participants affected / at risk) | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66
Other Adverse Events (participants affected / at risk) | 5/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm (N=66)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators are required to submit any proposed publications to the study sponsor for review and approval at least 60 days prior to submitting the materials for external publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT03417466/SAP_000.pdf
  • Study Protocol (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT03417466/Prot_001.pdf